CLINICAL TRIAL: NCT05962281
Title: Investigation The Effect of Conventional Vs. Individualized Transcranial Direct Current Stimulation Intensity to Achieve Uniform E-Fields
Brief Title: Investigation The Effect of Conventional Vs. Individualized tDCS Intensity to Achieve Uniform E-Fields
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Koen Cuypers (Other)
Collaborators: BOF-BILA (Unknown)
Responsible Party: Sponsor-Investigator, Koen Cuypers, Assoc. Prof., Hasselt University
Organization: Hasselt University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: B1152023000005; BOF23DOCBL02 (Other Grant/Funding Number: Special Research Fund (BOF))
Record Dates: First submitted 2023-06-02; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; Neurophysiologic Abnormality
Keywords: Multiple Sclerosis; Brain Stimulation; Non-invasive Brain Stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Individualized tDCS (Active Comparator): Each participant will be screened according to their brain scan, they will receive individualized dose of tDCS currents.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Fixed currents tDCS (Active Comparator): All of the participant will receive standardized dose of tDCS currents intensity of 2 mA.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): The electrodes will applied to the cortical areas, however none of all of the participant will receive the current dose of tDCS.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS), a form of non-invasive brain stimulation which involves the use of low intensity currents propagated via the scalp, is widely implemented as both a fundamental and clinical neuroscientific tool. Over the last decades, tDCS showed significant therapeutic promise, as numerous studies revealed that it can result in improved attention and executive functions in patients with neurological disorders, through modification of neuronal excitability.

SUMMARY:
Background: Replications of studies employing transcranial direct stimulation (tDCS) shows great variations in physiological and behavioral outcomes. The disparity between studies is based on the expectations of getting the same cortical activity changes consistently once the procedures and current parameters have been repeated. Nevertheless, this assumption was inoperative, due to the individualized variations of numerous parameters such as: age, disease type, symptom severity, head geometry, etc.

Objective: Through this clinical trial we aim to reduce the variability of the physiological and behavioral outcomes of tDCS by individualizing the current intensity and to study the neurophysiological and behavioral outcome differences between participants who receive the customized current intensity in comparison to the others who would receive a fixed dose.

Methods: Based on individual patient's structural MRI images, the Electrical field (E-field) distribution can be modeled and the individualized current dose to stimulate a target region can be determined. A group of thirty persons with multiple sclerosis (PWMS) would be pseudo-randomized into three groups receiving all 3 treatments of individualized tDCS, fixed currents (2 mA), and sham tDCS. Baseline and post-intervention assessment of physiological and behavioral outcome measures will be assessed using respectively, transcranial magnetic stimulation (TMS) recruitment curve and a stop-signal task and GO/No-go test.

Significant statement and clinical relevance: Individualizing the patient's tDCS current intensity will result in a better clinical outcome (i.e. more robust physiological and behavioral effects), as compared to a tDCS application that is based on a fixed current.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed volunteers, assessed by Edinburgh handedness inventory
* Normal or corrected-to-normal vision
* Greater than or equal to 18 years old
* Relapsing-remitting type of MS (RRMS)
* Moderate disability EDSS score ≤ 6.5
* Free of relapsing attack at least a month before recruitment

Exclusion Criteria:

* Subject recently had a seizure or epilepsy
* Subject is a habitual smoker;
* Subject has a history of any major disease that may interfere with the investigations (especially liver and kidney disease, upper limb pathologies, history of significant multiple traumas, or diabetes) or cancer;
* Subject has any history of a major neurological disorder in addition to MS (including previous severe brain trauma and cognitive impairment) or known cerebral structural abnormalities;
* Subject has a diagnosed mental disorder (e.g., depression, bipolar disorder, schizophrenia, psychoses);
* Subject is currently a user (including ''recreational use'') of any illicit drugs or has a history of drug or alcohol abuse;
* Subject has significant abnormalities on T1/T2 MRI scan;
* Subject has a contra-indication for MRI scanning or TMS measurements (see screening forms for MRI and TMS);
* Subject does not understand the study procedure;
* Subject is unwilling or unable to perform all study procedures, or is considered unsuitable in any way by the principal investigator;
* Subject is not able to perform the motor tasks;
* Subject is (potentially) pregnant (in case of doubt, hCG test will be conducted in female participants); subject is breastfeeding at the time of the study;
* Subject chronically uses medication, especially sedatives or sleep medication (contraceptives allowed). Other medication that is only taken as needed will be allowed at the investigator's discretion;
* Using TMS, no (sufficiently stable) MEPs can be evoked at left M1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) Assessment | Baseline assessment before tDCS session (Pre-intervention), and immediately following tDCS session (Post-intervention).
  Changes in cortical excitability will be measured by single and paired TMS pulses.
  The final values will be assessed for improvements.

SECONDARY OUTCOMES:
Behavioral Assessment | Baseline assessment before tDCS session (Pre-intervention), and immediately following tDCS session (Post-intervention).
  A cognitive test battery consisting of:
  1- Symbol Digit Modality Test (SDMT); the final score is the correct number of substitutions in 90 seconds, and scores range between 0 and 110, where higher scores indicating better outcome, and the lower scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Cuypers, PhD, Principal Investigator — UHasselt

IPD SHARING:
Plan to Share IPD: No